CLINICAL TRIAL: NCT05074862
Title: Effects of Ketosis on Muscle Kinetics and Signaling During Critical Illness.
Acronym: KETO-ICU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Berg-Hansen, MD, Principal Investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KETO-ICU 1-10-72-231-21
Record Dates: First submitted 2021-09-17; First posted 2021-10-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Intensive Care Unit Acquired Weakness; Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: A randomized double-blind isocaloric placebo-controlled cross-over study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone monoester (3-OHB) (Experimental): Weight-adjusted dose of 3-OHB Monoester (KetoneAID KE4, Virginia, US). Bolus of 300 mg/kg followed by a 2-hour continuous enteral infusion with a dosing of 100 mg/kg/hour (maximal total dose 50 grams). There is a 1-hour lag between the bolus and the continuous infusion.
  Interventions: Dietary Supplement: KetoneAid KE4 Pro Monoester
- Placebo Treatment (Placebo Comparator): Maltodextrin- and fatbased placebo in isocaloric, isovolemic dose to the experimental arm.
  Interventions: Dietary Supplement: Maltodextrin and fat-based placebo

INTERVENTIONS:
Dietary Supplement: KetoneAid KE4 Pro Monoester — A dietary supplement containing ketone monoester.
  Arms: Ketone monoester (3-OHB)
Dietary Supplement: Maltodextrin and fat-based placebo — Dosis isocaloric to the KetoneAid Arm
  Arms: Placebo Treatment

SUMMARY:
Background:

Patients with critical illness in the intensive care unit (ICU) experience marked skeletal muscle weakness, muscle atrophy and disability in physical function, commonly termed ICU-acquired weakness (ICU-AW). The pathophysiology of ICU-AW is complex, but a key feature of skeletal muscle wasting is disturbed protein metabolism reflected in both increased rate of muscle protein degradation and reduced synthesis. Treatment with 3-OHB seems a promising new anticatabolic treatment in patients with critical illness, preventing ICU-AW. To date, no data exist on the clinical and functional effects of ketone body modulation in patients with critical illness.

Objective:

The aim to investigate the effect of exogenous 3-OHB administration on muscle protein kinetics and lipolysis in patients with critical illness, aiming towards preventing ICU-AW.

Design:

A randomized double-blind isocaloric placebo-controlled cross-over study in 10 mechanically ventilated patients with critical illness in the ICU.

Methods:

Evaluation of whole-body and focal leg protein kinetics using labeled phenylalanine and tyrosine tracers. Assessment of free fatty acid (FFA) turnover using a labeled palmitate tracer. Femoral arterial blood flow (assessed with pulsed-wave Doppler ultrasound) is evaluated once per study period. Blood- and urinary samples are collected routinely throughout the study day. Whenever feasible, muscle and fat biopsies will be taken for analysis of protein and adipocyte metabolic signaling and mitochondrial function.

Perspectives: This investigation may grant essential knowledge on ketosis in critical illness. This may lead to larger clinical trials, and hopefully a new and better treatment strategy aimed at preserving muscle mass and function during and improving recovery after critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation via a cuffed endotracheal or tracheotomy tube.
* Expected survival of ICU admission.
* Adults (≥18 years).
* Multi-organ failure (Sequential Organ Failure Assessment Score [SOFA] score ≥2 in 2 or more domains).

Exclusion Criteria:

* Moribund or expected withholding treatment within 48 hours as judged by the investigator.
* Palliative goals of care.
* Contraindication for enteral nutrition.
* Pregnancy.
* Known severe musculoskeletal or neurological disability.
* Diabetic ketoacidosis.
* Phenylketonuria.
* BMI ≤17 or deemed malnourished as judged by the investigator.
* BMI >40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Net leg phenylalanine release | 3 hours
  As measured by rate of phenylalanine appearance in relation with the rate of disappearance.

SECONDARY OUTCOMES:
Change in rate of appearance of phenylalanine over the leg. | 3 hours.
Change in rate of disappearance of phenylalanine over the leg. | 3 hours.
Whole body palmitate flux | 3 hours.
  As measured by rate of appearance of a palmitate-tracer
Change in arterial pH. | 3 hours.
Changes in inflammatory cytokines (IL-1, IL-6, IL-18, TNFa) | 3 hours.
Changes in intramyocellular protein metabolic signalling pathways. | 3 hours.
  The Akt-, mTor-, and ubiquitin-proteasome pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No